CLINICAL TRIAL: NCT06406010
Title: A Blinded Randomized Study Investigating the Effect of Pericapsular Nerve Group (PENG) Block on Postoperative Pain After Peri-acetabular Osteotomy
Brief Title: Investigating the Effect of Pericapsular Nerve Group (PENG) Block on Postoperative Pain After Peri-acetabular Osteotomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, MD PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PENG for PAO
Record Dates: First submitted 2024-04-30; First posted 2024-05-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine group (Experimental): Ropivacaine 5 mg/ml 20ml
  Interventions: Drug: Ropivacaine 5mg/ml 20ml
- Saline group (Placebo Comparator): NaCl 0.9%
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Ropivacaine 5mg/ml 20ml — administered in a pericapsular nerve group (PENG) block
  Arms: Ropivacaine group
Drug: Saline 0.9% — administered in a pericapsular nerve group (PENG) block
  Arms: Saline group

SUMMARY:
The aim of this study is to determine the effect of PENG blockade on postoperative pain after either ropivacaine 5 mg/mL or saline (placebo) in patients undergoing PAO. The hypothesis of this study is that PENG block with ropivacaine reduces postoperative pain compared to placebo (saline).

DETAILED DESCRIPTION:
Peri-acetabular osteotomy (PAO) is the joint-preserving treatment of choice in young adults with symptomatic hip dysplasia. However, moderate to severe pain occurs frequently in the postoperative period. Pain after PAO comes primarily from the anterior hip capsule which is innervated by the terminal nerves of the lumbar plexus comprising branches from the femoral, obturator and accessory obturator nerves. The articular branches from the femoral nerve reach the plane between the iliopsoas muscle and the iliofemoral ligament (iliopsoas plane) and innervate the anterior and lateral aspects of the hip capsule. The articular branches innervate the anterior and medial aspects of the hip capsule and the accessory obturator nerve contributes to the innervation of the hip in 10%-30% of the patients, and supplies the inferomedial aspect of the hip capsule. The PAO procedure, involving three osteotomies in otherwise healthy individuals, is likely to produce a substantial surgical stress response, which potentially could be alleviated by multimodal analgesia including the pericapsular nerve group (PENG) block.

The PENG block is a novel regional anaesthesia technique that has been proposed as an effective motor-sparing block for total hip arthroplasty. The PENG block targets the articular branches providing innervation to the anterior capsule of the hip joint, including the femoral, obturator and accessory obturator nerves. Its potential analgesic and motor-sparing effect is desirable for early ambulation, better physical therapy, and earlier discharge.

Conventional opioid-sparing regional anaesthetic techniques such as lumbar plexus and femoral nerve blocks are effective but carry a risk of undesirable lower limb muscle weakness. Alternatively, the fascia iliaca block does not consistently provide adequate pain relief for hip surgeries.

The anterior capsule of the hip has a high density of nociceptors and mechanoreceptors and appears to be the primary source of pain after hip surgery. The PENG block targets the articular branches providing innervation to the anterior capsule of the hip joint, including the femoral, obturator and accessory obturator nerves.

A recent study reported improved quality of recovery and reduced opioid requirements for patients undergoing primary THA whereas other studies have reported conflicting results regarding the analgesic efficacy for THA. However, the effect of PENG on PAO has not been investigated.

Thus, in order to investigate if PENG block is superior to placebo in decreasing immediate pain and other complications after PAO, the investigators aim to conduct a randomised, double-blinded trial of ropivacaine 5 mg/ml vs. placebo. The investigators hypothesize that patients given ropivacaine 5 mg/ml will have less pain in the first 24 postoperative hours compared with patients given placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Informed consent
3. Scheduled for periacetabular osteotomy under general anesthesia with intubation
4. American Society of Anesthesiologists (ASA) physical status classification I to III
5. Can read and understand Danish

Exclusion Criteria:

1. Known allergy to ropivacaine
2. Daily use of opioids, gabapentin or tricyclic antidepressant (regardless of dose) within the last four weeks prior to surgery
3. Contraindications to Celocoxib, NSAIDs or paracetamol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain during first 24 hours postoperatively | 24 hours postoperatively
  Area under curve (AUC) of pain reported on a numeric rating scale (NRS) from 0 to 10 (where 0 is no pain and 10 is the worst pain imaginable) during the first 24 hours postoperatively

SECONDARY OUTCOMES:
Presence of moderate to severe pain | within 3 hours
  The number of patients reporting moderate to severe pain at rest [>3 out of 10 on a numeric rating scale (NRS) from 0 to 10 (where 0 is no pain and 10 is the worst pain imaginable)] at any point in the immediate postoperative phase (from arrival at the PACU until transfer to the ward). NRS will be assessed upon arrival at the PACU and each 30 minutes.
Pain during mobilization | within 5 hours
  Pain during during mobilization (from laying down in bed till standing on the floor) assessed on numeric rating scale (NRS) from 0 to 10 (where 0 is no pain and 10 is the worst pain imaginable) at 5 hours after extubation
Opioid use 24 hours | 24 hours
  Opioid use from tracheal extubation until 24 hours postoperatively
Pain during mobilization | within 24 hours
  Pain during during mobilization (from laying down in bed till standing on the floor) assessed on numeric rating scale (NRS) from 0 to 10 (where 0 is no pain and 10 is the worst pain imaginable) at:
  * postoperative day one between 8 and 10 pm
  * 24 hours after extubation
First opioid | within 24 hours
  Time to first opioid
Last opioid | within a week
  Time to last opioid
Time to first PONV-medication | within 24 hours
  Time to first PONV-medication
Opioid use at PACU | within 24 hours
  Opioid use at PACU
Sleep quality/pain during sleep. | within 24 hours
  During the first postoperative night the patients answer yes/no to whether they awoke from their sleep because of pain.
Length of stay at hospital | within a week
  Length of stay at hospital
Length of time to fulfilling PACU discharge criteria | within 24 hours
  Length of time to fulfilling PACU discharge criteria
Defecation | within 24 hours
  Time to first defecation

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, Md, PhD, Study Chair — Rigshospitalet University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No